CLINICAL TRIAL: NCT02652715
Title: A Pilot Feasibility Trial of the Tolerability of Oral Salvia Hispanica and Its Effect on Blood Fatty Acids and Stool Microbiome in Patients With Treated Non-Hodgkin Lymphoma
Brief Title: Salvia Hispanica Seed in Reducing Risk of Disease Recurrence in Patients With Non-Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LS1581; NCI-2015-02149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-006720; LS1581 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-01

CONDITIONS: Adult Nasal Type Extranodal NK/T-Cell Lymphoma; Adult T-Cell Leukemia/Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma; B Lymphoblastic Leukemia/Lymphoma; Blastic Plasmacytoid Dendritic Cell Neoplasm; Burkitt Leukemia; Central Nervous System Lymphoma; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Diffuse Large B-Cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3 Follicular Lymphoma; Hepatosplenic T-Cell Lymphoma; Lymphoplasmacytic Lymphoma; Mantle Cell Lymphoma; Mediastinal (Thymic) Large B-Cell Lymphoma; Mycosis Fungoides; Nasal Type Extranodal NK/T-Cell Lymphoma; Nodal Marginal Zone Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Post-Transplant Lymphoproliferative Disorder; Primary Cutaneous Anaplastic Large Cell Lymphoma; Primary Effusion Lymphoma; Sezary Syndrome; Splenic Marginal Zone Lymphoma; Subcutaneous Panniculitis-Like T-Cell Lymphoma; Systemic Anaplastic Large Cell Lymphoma; T Lymphoblastic Leukemia/Lymphoma; Transformed Recurrent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma; Blastic Plasmacytoid Dendritic Cell Neoplasm; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Lymphoma, T-Cell; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Lymphoma, Primary Effusion; Sezary Syndrome; Subcutaneous panniculitis-like T-cell lymphoma | interventions — Salvia hispanica seed extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Basic science (Salvia hispanica seed) (Experimental): Patients receive Salvia hispanica seed PO QD for 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Dietary Supplement: Salvia hispanica Seed

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Dietary Supplement: Salvia hispanica Seed — Given PO
  Other Names: Chia; Chia Seed; SH Seed

SUMMARY:
This pilot clinical trial studies Salvia hispanica seed in reducing the risk of returning disease (recurrence) in patients with non-Hodgkin lymphoma. Functional foods, such as Salvia hispanica seed, has health benefits beyond basic nutrition by reducing disease risk and promoting optimal health. Salvia hispanica seed contains essential poly-unsaturated fatty acids, including omega 3 alpha linoleic acid and omega 6 linoleic acid; it also contains high levels of antioxidants and dietary soluble fiber. Salvia hispanica seed may raise omega-3 levels in the blood and/or change the bacterial populations that live in the digestive system and reduce the risk of disease recurrence in patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess if dietary supplementation with the functional food Salvia hispanica (SH) seed improves serum omega-3 (n-3) fatty acids (FA) levels in patients with non-Hodgkin lymphoma (NHL) who have recently completed chemotherapy.

SECONDARY OBJECTIVES:

I. Evaluate the safety and tolerability of patients taking 16 grams (g) (approximately 1 United States [US] tablespoon) of SH per day.

II. Evaluate the compliance of stool sample collection in lymphoma patients who have completed therapy and are in remission.

III. Evaluate if SH can exert measurable changes of the stool microbiome. IV. Evaluate if changes in n-3 levels and stool microbiome persist or resolve after participants are no longer taking SH.

OUTLINE:

Patients receive Salvia hispanica seed orally (PO) once daily (QD) for 12 weeks.

After completion of study, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of any type of NHL and =< 5 years from the last treatment
* In remission (complete remission [CR], partial remission [PR], or stable disease based on clinical, not necessarily radiologic, assessment) and currently being observed and with no current cytotoxic chemotherapy planned; patients may be on rituximab maintenance
* No international travel planned during the next 4 months
* Able to eat a full range of solid food and liquids and tolerate seeds/nuts
* Maintain a consistent general diet without significant variation
* Able to deliver four fresh (within 24 hours) stool samples to Mayo Clinic Rochester over a four month period
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Provide informed written consent
* Able to recollect dietary intake for the prior 24 hours in order to complete a one-day food record with assistance from a dietician at each study visit
* Willing to complete the food frequency questionnaire (FFQ) at baseline and at 16 week visits with assistance from a dietician
* Willing to be seen at baseline, 6 weeks, 12 weeks, and 16 weeks for the study time points
* Willing to provide blood and stool samples at baseline and study time points for correlative research purposes

Exclusion Criteria:

* Cannot eat normal table food by mouth; NOTE: patients with any form of feeding tube or a swallowing disorder are not eligible
* Have taken fish oil, another dedicated n-3 supplement, or SH seed from another source within the last 28 days; patients on multivitamins that contain n-3 are eligible
* Co-morbid systemic illnesses such as active infection or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens; NOTE: patients with significant gut malabsorptive conditions (such as inflammatory bowel disease or others at the discretion of the investigator) will be excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent that would be considered as a treatment for the lymphoma; NOTE: rituximab maintenance and patients participating on Mayo Clinic vitamin D study are allowed
* Active other malignancy requiring treatment that would interfere with the assessments of this study
* Major surgery other than diagnostic surgery =< 4 weeks prior to registration
* On prophylactic antibiotics, such as trimethoprim-sulfamethoxazole for pneumocystis prophylaxis or post-transplant penicillin prophylaxis
* Have taken antibiotics =< 7 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Changes in improvement of n-3 serum alpha-linoleic acid levels | Baseline to up to 16 weeks
  n-3 level will be evaluated as a continuous measure, where the median and range will be summarized at each time point. Changes across time will be evaluated graphically. Changes from baseline will be quantitatively summarized and will be evaluated using paired sample methods (paired sample t-test).

SECONDARY OUTCOMES:
Changes in n-3 levels after participants are no longer taking SH | From 12 weeks to up to 16 weeks
  The evaluation of whether changes in n-3 levels persist or resolve after participants are no longer taking SH will be assessed using a paired t test comparing the mean values at 12 weeks to the mean values at 16 weeks. Changes from week 12 to week 16 will also be calculated and the mean magnitude of change will be explored.
Changes in stool microbiome after participants are no longer taking SH | From 12 weeks to up to 16 weeks
  The evaluation of whether changes in stool microbiome persist or resolve after participants are no longer taking SH will be assessed using a paired t test comparing the mean values at 12 weeks to the mean values at 16 weeks. Changes from week 12 to week 16 will also be calculated and the mean magnitude of change will be explored.
Changes in stool microbiome after supplementation with SH, assessed by gene sequencing | Baseline to up to 16 weeks
  Patient's initial sample will provide a control to assess alterations in stool deoxyribonucleic acid (DNA) (reflecting stool bacterial populations) after supplementation with SH. Measurable change will be assessed based on standardized methods.
Incidence of adverse events graded according to the National Cancer Institute Common Toxicity Criteria version 4.0 | Up to 16 weeks
  Safety and tolerability will be assessed utilizing stool and symptom diaries. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. The relationship of the adverse event(s) to the study treatment will be taken into consideration. In addition, tolerability will be further assessed by evaluating the number of doses missed due to adverse events. Reasons for missed doses will be summarized.
Patient compliance in stool sample collection | Up to 16 weeks
  Patient compliance in stool sample collection will be assessed by evaluating the percentage of patients who provide a sample at each time point. The percentage of patients who provide samples for 0, 1, 2, 3, or all 4 time points will be calculated to determine the feasibility of requesting multiple samples on future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Witzig, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States